CLINICAL TRIAL: NCT06508190
Title: Impact of Free Walking Exercise on Obstructive Sleep Apnea Patients With Non-alcoholic Fatty Liver on Liver Enzymes, Degree of Exhaustion, and Quality of Sleep
Brief Title: Free Walking Exercise in Obstructive Sleep Apnea Patients With Non-alcoholic Fatty Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed El-Hadidy, lecturer, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03202405263221
Record Dates: First submitted 2024-07-13; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea; Non-alcoholic Fatty Liver
MeSH Terms: conditions — Sleep Apnea, Obstructive; Non-alcoholic Fatty Liver Disease | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Forty patients suffering from obstructive sleep apnea are divided into two groups: one for CPAP and the other for CPAP and free walking program.
Who Masked: Outcomes Assessor
Masking Description: The authors of this clinical trial and patients do not provide the study outcome examiners with information regarding device therapy or free walking exercise.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous positive airway pressure therapy (Active Comparator): The continuous positive airway pressure therapy equipment is used for 12 weeks, all patients in this group groups must utilize the CPAP machine for 4 hours each night.
  Interventions: Behavioral: continuous positive airway pressure
- Free walking & continuous positive airway pressure therapy (Experimental): Each patient is required to walk 30 minutes, seven days a week for 12 weeks.
  & The continuous positive airway pressure therapy equipment is used for 12 weeks, all patients in both groups must utilize the CPAP machine for 4 hours each night.
  Interventions: Behavioral: free walking exercise and continuous positive airway pressure

INTERVENTIONS:
Behavioral: continuous positive airway pressure — continuous positive airway pressure therapy for a period of 12 weeks, all patients with in this group are required to utilize the CPAP machine for at least 4 hours each night
  Arms: continuous positive airway pressure therapy
Behavioral: free walking exercise and continuous positive airway pressure — patients will receive continuous positive airway pressure therapy for a period of 12 weeks, all patients with in this group are required to utilize the CPAP machine for at least 4 hours each night. Also, patients will perform walking exercise for 30 mint, daily for 12 weeks
  Arms: Free walking & continuous positive airway pressure therapy

SUMMARY:
Research evaluating the impact of continuous positive airway pressure (CPAP) & walking exercise on fatigue severity, liver enzymes and sleeping quality in patients with non-alcoholic fatty liver disease who also have obstructive sleep apnea. Forty patients are divided into two groups: twenty patients CPAP and other twenty patients for CPAP and walking program .

DETAILED DESCRIPTION:
Research evaluating the impact of continuous positive airway pressure (CPAP) & walking exercise on fatigue severity, liver enzymes and sleeping quality in patients with non-alcoholic fatty liver disease who also have obstructive sleep apnea. Forty patients are divided into two groups: twenty patients CPAP and other twenty patients for CPAP and walking program .

ELIGIBILITY:
Inclusion Criteria:

* The body mass index (BMI) < 35 kg/m2.
* obstructive sleep apnea patients with fatty liver

Exclusion Criteria:

* liver transplantation , alcoholic fatty liver, antipsychotic medications, bariatric surgery; cardiac , renal problem , liver cancer ; pregnancy,orthopedic problems, systemic diseases, respiratory dysfunctions, neurological dysfunctions.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Alanine tranaminase | it will be measured after 12 weeks
  serum hepatic enzyme

SECONDARY OUTCOMES:
Asparatate transamianse | it will be measured after 12 weeks
  serum hepatic enzyme
Body mass index | it will be measured after 12 weeks
  it will be masusured on empty stomach and bladder
triglycerodes | it will be assessed after 12 weeks
  it will be meausred in plasma
Pittsiburg sleeping quality index | it will be assessed after 12 weeks
  a questionnaire that wil be used for assessing sleeping quality
fatigue severity scale | it will be assessed after 12 weeks
  a questionnaire that wil be used for assessing fatigue
Epworth sleepness scale | it will be assessed after 12 weeks
  a questionnaire that wil be used for daytime sleepness

CONTACTS AND LOCATIONS:
Overall Officials: El-Hadidy Hagar, Principal Investigator — Faculty of Physical Therapy, Ahram Canadian University (ACU), Giza, Egypt
Locations (1):
- Ahram canadian university, Giza, Egypt